CLINICAL TRIAL: NCT04982900
Title: A Prospective, Multi-center, Double-blind Randomized Controlled Clinical Trial on the Treatment of EGFR-TKI for Residual Lesions of Multiple Synchronous Ground-glass Opacities
Brief Title: Treatment of EGFR-TKI for Residual Lesions of Multiple Synchronous Ground-glass Opacities
Acronym: TERMGGO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Tang-Du Hospital (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTS-015
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Multiple Primary Lung Cancers
Keywords: Multiple Primary Lung Cancer; Ground-glass Opacity; EGFR-TKI; Targeted Therapy
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Intervention Model Description: This study has two parallel arms, EGFR-TKI treatment arm and control arm (placebo) are included in this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind trial, the investigator, care provider and patients are all blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGFR-TKI Treatment Arm (Experimental): After randomization, the enrolled patients in this arm should be completely free from the risk of perioperative complications or recovered from the effects of complications, usually no earlier than 4 weeks after surgery but no more than 10 weeks after surgery, before receiving baseline follow-up and starting oral administration of Furmonertinib on the day of baseline follow-up. Patients in the treatment group should take Furmonertinib (80 mg each time) orally on an empty stomach before breakfast once a day. The medicine should be taken about the same time each day, by swallowing the whole tablet with water, without crushing or chewing. Patients should maintain oral administration of Furmonertinib for 6 consecutive months, unless there is disease progression, death, new anti-tumor therapy received or intolerance of investigational drugs.
  Interventions: Drug: furmonertinib
- Control Arm (Placebo Comparator): After randomization, the enrolled patients in this arm should be completely free from the risk of perioperative complications or recovered from the effects of complications, usually no earlier than 4 weeks after surgery but no more than 10 weeks after surgery, before receiving baseline follow-up and starting oral administration of placebo on the day of baseline follow-up. Patients in the treatment group should take placebo (80 mg each time) orally on an empty stomach before breakfast once a day. The medicine should be taken about the same time each day, by swallowing the whole tablet with water, without crushing or chewing. Patients should maintain oral administration of placebo for 6 consecutive months, unless there is disease progression, death, new anti-tumor therapy received or intolerance of investigational drugs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: furmonertinib — AST2818 is an irreversible and highly selective EGFR inhibitor independently discovered and developed by Allist. It has the potential to become the best-in-class drug in the third-generation EGFR-TKIs. Data from the preclinical studies and the completed clinical studies show that AST2818 has the following advantages: 1) AST2818 has good target selectivity and tissue distribution specificity; 2) The objective response rate of AST2818 for the patients with locally advanced or metastatic NSCLC with EGFR T790M mutation is outstanding, reaching 74.1% in the key registration clinical study; 3) AST2818 has a good safety profile and is well-tolerated; 4) AST2818 and its active metabolites have a superior ability to penetrate the blood-brain barrier, and have a good therapeutic efficacy on brain metastases frequently seen in patients with NSCLC.
  Other Names: AST2818
  Arms: EGFR-TKI Treatment Arm
Drug: Placebo — The placebo has the same appearance, weight, and physical and chemical properties as the study drug, and is provided by the researcher to the subjects in control group.
  Arms: Control Arm

SUMMARY:
This study is a multi-center, prospective, double-blind randomized controlled clinical trial. The purpose is to evaluate the efficacy and safety of EGFR-TKI on residual GGOs after surgery in patients with multiple primary lung cancers with ground glass nodules. This study is expected to prove that compared with placebo in the control group, EGFR-TKI can significantly reduce the residual GGOs lesions in patients with EGFR-positive multiple primary lung cancers with ground-glass opacity, and bring a higher objective response rate (ORR), thus provides new insights for treatment of these patients.

DETAILED DESCRIPTION:
Lung cancer is one of the most deadly malignant tumors in the world. It is estimated that 0.2-20% of lung cancer patients have multiple primary lung cancers at the time of diagnosis, and many of them present with multiple ground glass opacities. The surgical method for such multiple lesions depends on their number, anatomical location and size, as well as the age and pulmonary function of the patient. It is easily affected by the subjective judgment of the surgeon. Besides, many of these patients develop multiple lesions that cannot be resected at the same time, and there haven't been established a standard therapy for residual GGO lesions after surgery.

According to the National Comprehensive Cancer Network (NCCN) guidelines, EGFR-TKI is recommended for the adjuvant treatment of stage IB-ⅢA NSCLC with EGFR mutations. However, it is not clear whether EGFR-TKI is effective for multiple primary lung cancers or the residual GGOs after surgical resection of the EGFR mutation positive main cancers. At present, there have been retrospective studies showing that application of EGFR-TKIs targeted therapy can significantly reduce the diameter of residual GGOs after surgery resection of EGFR mutation-positive primary lesions for MPLC patients, and reduce the secondary surgery caused by the progression of the lesion. However, there is no prospective Studies confirming the efficacy and safety of EGFR-TKI on these postoperative residual GGOs lesions.

This study is a multi-center, prospective, double-blind, comparative clinical research. This study plans to enroll 138 patients with multiple primary lung cancers (cTis-T1c, N0, M0) that manifest GGO and cannot be resected at the same time, patients should have undergone surgical resection of the EGFR mutated main lesion, and have no less than 1 GGO lesion remaining after surgery. Eligible patients will be randomly divided into the treatment group (receiving furmonertinib mesilate tablets) or control group (placebo) at a ratio of 1:1. The grouping process was strictly double-blind for both the investigators and subjects. By collecting the relevant data of patients' baseline images, pathology, and follow-up images during treatment, statistical analysis is used to evaluate the effectiveness (response rate, objective remission rate), safety, and relevant influencing factors (including CTR value of the main lesion, number of residual lesions, diameter of the largest residual lesion, higher stage of the main lesion, residual lesion's density, etc.) of EGFR-TKI treatment.

This study is expected to prove that compared with the placebo in the control group, EGFR-TKI can significantly reduce the diameter of residual GGO lesions in patients with EGFR-positive multiple primary lung cancers with ground-glass density, and bring a higher objective response rate (ORR) but did not significantly increase the incidence of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient was diagnosed with MPLC (based on the previously published MM/ACCP clinical criteria). The preoperative chest CT scan (1mm slice thickness) found two or more ground glass lesions (≥6mm and <3 cm, pure ground glass or partial solid) that could not be operated at the same time;
* 2. The patient has received surgery to remove the main lesion. The pathology of the main lesion is NSCLC with sensitizing EGFR mutation positive (19del/L858R), with or without other EGFR mutations including T790M;
* 3. After resection of the main lesion, the patient should have at least one residual ground glass nodules (≥6mm and <3 cm) that are suspected of being malignant and cannot be resected simultaneously with main lesion. The malignancy has been confirmed by both qualified radiologist and thoracic surgeon;
* 4. The included MPLC patients' clinical staging from preoperative evaluation should be cTis-T1c, N0, M0 (according to NCCN/EEJC 2021 V1);
* 5. Patients' ECOG PS score 0-1;
* 6. The subject voluntarily participates in the study and has signed a written informed consent form.

Exclusion Criteria:

* 1. MPLC with lymph node metastasis, unresectable disease or distant metastasis, including pleural and pericardial metastasis;
* 2. Those who have severe cardiac, pulmonary, hepatic, and renal failure and cannot tolerate surgery;
* 3. Patients suffering from other malignant tumors or a history of other malignant tumors within 5 years; except effectively controlled skin basal cell carcinoma, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, superficial bladder tumor, etc.;
* 4. Patients requiring long-term use of strong CYP3A4 inhibitors or strong inducers within 7 days before the first administration or during the expected test period;
* 5. Patients who are receiving medications that are known to prolong the QTc interval or may cause torsade de pointes ventricular tachycardia, and who need to continue to receive these medications during the study period;
* 6. History of interstitial lung disease (ILD), or drug-induced interstitial lung disease;
* 7. Severe gastrointestinal dysfunction, diseases or clinical conditions that may affect the intake, transport or absorption of the study drug, such as inability to take the drug orally, uncontrollable nausea and vomiting, history of extensive gastrointestinal resection, uncured recurrent diarrhea, atrophic gastritis (onset age less than 60 years old), uncured gastric diseases requiring proton pump inhibitors (omeprazole, lansoprazole, pantoprazole, raneprazole, etc.) , Crohn's disease, ulcerative colitis, etc.;
* 8. Cardiovascular diseases which meet any of the following: (1) In the resting state, the QTc interval of ECG is >470 msec; (2) Severe abnormalities in heart rhythm, cardiac conduction, and resting ECG, such as complete left bundle branch block, third degree heart block, second degree heart block, PR interval> 250 msec, etc.; (3) Any factors that may increase the risk of QTc interval prolongation or the risk of arrhythmia events, such as heart failure, hypokalemia, hypomagnesemia, etc., congenital long QT syndrome, family history of long QT syndrome, Sudden death unexplained in first-degree relatives under 40 years of age or use of any drug combination that is known to prolong the QTc interval and cause torsion de pointes tachycardia; (4) Left ventricular ejection fraction (LVEF) <50%; (5) Having a history of myocardial infarction, severe or unstable angina, or coronary artery bypass surgery in the last 6 months, or cardiac insufficiency grade ≥ NYHA grade 2; (6) Uncontrollable hypertension (systolic blood pressure ≥150mmHg and/or diastolic blood pressure ≥100mmHg);
* 9. Active period of infectious diseases, such as hepatitis B, hepatitis C and human immunodeficiency virus (HIV) infections;
* 10. Women who are pregnant or breastfeeding, or have fertility but have not taken contraceptive measures;
* 11. People who suffer from uncontrollable neurological or mental illnesses or mental disorders, having poor compliance, cannot cooperate or describe treatment responses;
* 12. Participants in other clinical trials at the same time or expect to receive other anti-tumor treatments outside of this study during the trial period;
* 13. Other situations that researchers think are not suitable for participating in this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Response rate of EGFR-TKI | 6 months
  defined in this study as the ratio of patients with reduced diameter of any residual lesions on CT scans to the entire patient cohort according to the Independent Review Committee (IRC) image evaluation follow-up.

SECONDARY OUTCOMES:
Lesion-oriented EGFR-TKI response rate | 6 months
  Defined as the ratio of lesions showing any reduction in diameter on the CT scan to the number of lesions in the entire cohort according to the Independent Review Committee (IRC) image evaluation during follow-up.
Objective response rate (ORR) | 6 months
  ORR is evaluated after 6 months of treatment, defined according to the RECIST1.1 standard
Response rate by Investigators' assessment | 6 months
  compared with the primary endpoint of Independent Review Committee (IRC) image evaluation
Second operations | 6 months
  Number of subjects who had a second resection of residual lesions due to progress of lesions during follow-up.
Treatment-related adverse events | 6 months
  the number and grades of treatment-related adverse events in each arm (grading according to CTCAE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, PhD, MD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (6):
- China (6):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No